CLINICAL TRIAL: NCT02179359
Title: MT2014-10C: Allogeneic Hematopoietic Stem Cell Transplant for Patients With High Risk Hemoglobinopathies and Other Red Cell Transfusion Dependent Disorders
Brief Title: Hematopoietic Stem Cell Transplant for High Risk Hemoglobinopathies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced by another study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014OC034; MT2014-10C (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease; Transfusion Dependent Alpha- or Beta- Thalassemia; Diamond Blackfan Anemia; Paroxysmal Nocturnal Hemoglobinuria; Glanzmann Thrombasthenia; Severe Congenital Neutropenia; Shwachman-Diamond Syndrome; Non-Malignant Hematologic Disorders
Keywords: Stem Cell Transplant
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; Anemia, Diamond-Blackfan; Hemoglobinuria, Paroxysmal; Thrombasthenia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Shwachman-Diamond Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Reduced Toxicity Ablative Regimen (Experimental): For use in patients with a matched sibling donor or unrelated UCB donor and DBA patients who are <12 years and/or have mild/moderate iron exposure.
  Interventions: Drug: Reduced Toxicity Ablative Regimen
- Reduced Intensity Preparative Regimen (Experimental): For use in patients with unrelated donor bone marrow and for DBA patients who are >12 years and/or have significant iron exposure.
  Interventions: Drug: Reduced Intensity Preparative Regimen
- Myeloablative Preparative Regimen (Experimental): For use in patients with a matched sibling donor, unrelated umbilical cord blood and in those with severe thalassemia.
  Interventions: Drug: Myeloablative Preparative Regimen

INTERVENTIONS:
Drug: Reduced Toxicity Ablative Regimen — * Anti-thymocyte Globulin (ATG)
  * Fludarabine
  * Busulfan
  * Stem Cell Infusion Day 0
  Arms: Reduced Toxicity Ablative Regimen
Drug: Reduced Intensity Preparative Regimen — * Alemtuzumab
  * Cyclophosphamide
  * Fludarabine
  * Total Body Irradiation (TBI)
  * Stem Cell Infusion Day 0
  Arms: Reduced Intensity Preparative Regimen
Drug: Myeloablative Preparative Regimen — * Alemtuzumab
  * Cyclophosphamide
  * Busulfan
  * Stem Cell Infusion Day 0
  Arms: Myeloablative Preparative Regimen

SUMMARY:
This is a study to collect the outcomes of stem cell transplantation for patients with hematologic diseases other than cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sickle Cell Disease, Thalassemia, Diamond Blackfan Anemia or other non-malignant hematologic disorders for which a stem cell transplant is indicated
* Acceptable stem cell source identified
* Performance status of ≥ 70% (Karnofsky),or ≥ 70 (Lansky play score)
* Creatinine <2.0 mg/dl for adults or glomerular filtration rate > 50 ml/min for children
* Bilirubin, Aspartate Aminotransferase, Alkaline phosphatase <5 times the upper limit of institutional normal
* Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction > 40%

Exclusion Criteria:

* active, uncontrolled infection
* pregnant or breastfeeding
* HIV positive

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09-02; Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
incidence of graft failure | 42 days

SECONDARY OUTCOMES:
overall survival | 6 months, 1 and 2 years
disease free survival | 6 months, 1 and 2 years
  patient no longer needing red blood cell transfusion and/or a hemoglobin S level at that of the donor ( sickle cell disease only)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Gupta, MBBS, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States